# Healthcare disparities in vitiligo: UK population-based cohort study

**Author names:** Viktoria Eleftheriadou<sup>1</sup>, Alia Ahmed<sup>2,3</sup>, John Nesnas<sup>4</sup>, Ranjit Nagra<sup>4</sup>

#### **Author affiliations:**

- $^{\rm 1}$  Department of Dermatology, The Royal Wolverhampton NHS Trust, Wolverhampton, UK
- <sup>2</sup> Frimley Health NHS Foundation Trust, Frimley, UK
- <sup>3</sup> Barts Health NHS Trust, London, UK
- <sup>4</sup> Pfizer Ltd, Walton Oaks, Walton on the Hill, Tadworth, Surrey, UK

**Date of the document:** August 25, 2023

# 1. Contents

| 1. | Cor | itent | S | 2 |
|---|---|---|---|---|
| 2. | List | of a | bbreviations | 4 |
| 3. | Inti | odu | ction | 5 |
| | 3.1 | Bac | kground | 5 |
| | 3.2 | Pur | pose of Analysis | 6 |
| 4. | Stu | dy ol | bjectives and endpoints | 6 |
| | 4.1 | Stu | dy Objectives | 6 |
| | 4.2 | Prii | mary Objectives | 6 |
| | 4.2 | .1 | Objective 1 | 6 |
| | 4.3 | Sec | ondary Objectives | 6 |
| | 4.3 | .1 | Objective 2 | 6 |
| | 4.3 | .2 | Objective 3 | 7 |
| | 4.3 | .3 | Objective 4 | 7 |
| | 4.3 | .4 | Objective 5 | 7 |
| | 4.4 | Pri | mary Endpoints | 7 |
| | 4.5 | Sec | ondary Endpoints | 7 |
| 5. | Ger | ieral | Study Design and Plan | 8 |
| | 5.1 | Stu | dy design | 8 |
| | 5.2 | Tot | al disease burden; cumulative lifetime risk | 8 |
| | 5.3<br>work | | parities in the impact of vitiligo on mental health, healthcare utilisation an | |
| | 5.4 | Dat | a Source and Read codes | 9 |
| | 5.5 | Dat | a Governance | 9 |
| | 5.6 | Dat | a Extraction | 9 |
| | 5.7 | Gen | neral Study Population | 9 |
| | 5.7 | .1 | Vitiligo Definition | 9 |
| | 5.7 | .2 | Sociodemographic subgroups1 | 0 |
| 6. | San | nple | Size Calculations1 | 0 |
| 7. | Pop | oulat | ions to be Analysed1 | 0 |
| | 7.1 | Incl | lusion Criteria1 | 0 |
| | 7.2 | Exc | lusion Criteria1 | 1 |
| | 7.3 | Mat | tching Process 1 | 1 |

| 8. | Stat | istical Analysis | .12 |
|-----|------|-----------------------------|-----|
| 8 | .1 | Statistical Principles | .12 |
| 8 | .2 | Primary Endpoint Analysis | .12 |
| 8 | .3 | Secondary Endpoint Analysis | .13 |
| 8 | .4 | Sensitivity Analysis | .14 |
| 8 | .5 | Missing Data | .14 |
| 9. | Stu | dy Limitations | .14 |
| 10. | Stat | cistical Software | .15 |
| 11. | Eth | ics | .15 |
| 12. | Ack | nowledgments | .16 |
| | | erences | |
| 14. | App | oendices | .18 |

# 2. List of abbreviations

| Abbreviation | Full Form |
|---|---|
| ADEPT | Anonymised Data Ethics & Protocol Committee |
| BMI | Body Mass Index |
| CIOMS | Council for International Organizations of Medical Sciences |
| EMA | European Medicines Agency |
| ENCePP | European Network of Centres for Pharmacoepidemiology and Pharmacovigilance |
| EQUATOR | Enhancing the QUAlity and Transparency Of health Research) |
| GEP | Good Epidemiological Practice |
| GP | General Practitioner |
| GPP | Guidelines for Good Pharmacoepidemiology Practices |
| IAPT | Improving Access to Psychological Therapies and psychiatric reviews |
| ICD10 | International Statistical Classification of Diseases and Related Health Problems 10th Revision |
| IEA | International Epidemiological Association |
| IMD | Index of Multiple Deprivation |
| IQR | Interquartile Range |
| ISPOR | International Society for Pharmacoeconomics and Outcomes<br>Research |
| OPCRD | Optimum Patient Care Research Database |
| SD | Standard Deviation |
| SES | Socio-Economic Status |
| SNOMED CT | Systemized Nomenclature of Medicine – Clinical Terms |
| UK | United Kingdom |

## 3. Introduction

## 3.1 Background

Vitiligo is an acquired, non-contagious skin disorder characterised by depigmented patches of skin that may appear in a localised or very generalised distribution, and affecting 0.5-2.0% of the global population.(1) The exact cause of the loss of functioning melanocytes in vitiligo remains unknown, but is likely to be resulted from the complex interplay of genetics, oxidative stress, and autoimmunity.(2)

Although vitiligo is typically asymptomatic, recent Pfizer-funded research has demonstrated the condition substantially affects psychological wellbeing.(3) This previous study showed that people with vitiligo have a considerable excess mental health burden when compared with people without vitiligo. It also showed that, in people with vitiligo, mental health comorbidity is associated with higher levels of healthcare utilisation, time off work, and unemployment.(3) This increased burden could be due to the unpredictable prognosis, the current lack of cure, the perception and emotional burden associated with the visibility of vitiligo, or a combination of these factors.

There is substantial scope to extend the initial analysis, with a comprehensive assessment of sociodemographic disparities in healthcare utilisation and in the burden of mental health comorbidity in people with vitiligo. Whilst the previous Pfizer-funded study demonstrated a difference by ethnicity in the mental health impacts of vitiligo (with vitiligo associated with a greater mental health burden in people of non-white ethnicity), the study was not designed to assess this as a primary outcome. Further analysis is required to fully understand these potential relationships as well as provide critical information on whether there is a socio-economic (SES) gradient in the mental health impacts of vitiligo. The previous study did not assess other potential disparities in management, such as healthcare utilisation of primary care encounters or dermatology services.

There is also substantial scope to expand on the previous study to provide, for the first time, a greater understanding of the total burden of vitiligo across the population, including reporting lifetime risk estimates for vitiligo, across sociodemographic groups. It is likely that substantial disease burden differences exist across these groups.

A comprehensive assessment of potential disparities in healthcare utilisation in vitiligo, mental health and social impact, and lifetime risk are needed. This research would both strongly complement previous Pfizer-funded work and support the use of newer therapies in vitiligo.

## 3.2 Purpose of Analysis

This study will provide the first estimate of the cumulative lifetime risk of vitiligo in the population overall, and by important sociodemographic groups, including age, sex, ethnicity and SES, which will prevalent key data to show the relative burden of vitiligo across the aforementioned groups. These approaches allow creation of cumulative lifetime risk plots which provide an excellent and accessible way to display the relative disease burden across groups.

This study will provide a detailed assessment of any sociodemographic disparities in comorbidities and social impact that occurs in people with vitiligo. This will include any differences in mental health impact of vitiligo by sociodemographic. It will also include a description of any sociodemographic disparities in time off work ("sick leave") or unemployment in people with vitiligo.

This study will also provide a detailed assessment of any sociodemographic disparities in healthcare utilisation in people with vitiligo with comparison across sociodemographic. This will include analysis of utilisation of primary care services, mental health referrals as well as referrals to secondary care (dermatology).

## 4. Study objectives and endpoints

## 4.1 Study Objectives

The overall purpose of the study is to provide an estimate of the lifetime risk of vitiligo in the population overall and by important sociodemographic groups. Moreover, to do a subgroup analysis in the vitiligo population to identify health-related disparities across people in different sex, age, deprivation and ethnicity.

## 4.2 Primary Objectives

## 4.2.1 Objective 1

Describe the total burden of vitiligo (cumulative lifetime risk) across sociodemographic subgroups.

## 4.3 Secondary Objectives

## 4.3.1 Objective 2

Describe any disparities in the burden of mental health outcomes, including depression and anxiety in people with vitiligo across sociodemographic subgroups.

## 4.3.2 Objective 3

Describe any disparities in the association of vitiligo with parasuicide/suicide attempts, adjustment disorder and sleep disturbances associated with vitiligo across sociodemographic subgroups.

## 4.3.3 Objective 4

Describe any disparities in vitiligo-associated healthcare utilisation across sociodemographic subgroups.

## 4.3.4 Objective 5

Describe any disparities in vitiligo-associated work impact (time off work for illness and unemployment) across sociodemographic subgroups.

## 4.4 Primary Endpoints

| Objective | Endpoints |
|---|---|
| 1 | An incident diagnosis of vitiligo is the date of the first diagnosis code in |
| | the record and no alternative diagnosis that merits exclusion (other |
| | causes of skin hypopigmentation) diagnosed within a one-year period (six |
| | months before or after their first vitiligo diagnosis code). |

Table 1: Primary endpoints.

## 4.5 Secondary Endpoints

| Objective | Endpoints |
|---|---|
| 2 | Mental health condition outcomes will be assessed up to two years post-<br>vitiligo diagnosis, including history of prior mental health condition and<br>will comprise of depression (record of any depressive episodes and/or<br>major recurrent depression diagnosis) and anxiety disorders, defined by<br>the International Statistical Classification of Diseases and Related Health<br>Problems 10th Revision (ICD10) classification, and identified using<br>algorithms validated for use in UK primary care data (See previously<br>published codes lists: (4)) |
| 3 | Other mental health condition outcomes will be assessed up to two years post-vitiligo diagnosis and will comprise of parasuicide/suicide attempts, adjustment disorder and sleep disturbance, defined by the International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD10) classification, and identified using algorithms validated for use in UK primary care data (See previously published codes lists: (4)) |

Healthcare utilisation outcomes will comprise primary care visits, dermatology referrals, mental health referrals (including but not limited to those via IAPT; Improving Access to Psychological Therapies and psychiatric reviews) in the two years post-vitiligo diagnosis.
 Unemployment in the two years post-vitiligo diagnosis will be identified using Read codes relating to unemployment recorded in the primary care record or the issuing of IB113 or ESA113 forms (See previously published codes lists: (4)).
 Time off work in the two years post-vitiligo diagnosis will be indicated by the issuing of Med 3 certification from primary care (Statement of Fitness for Work certification) (See previously published codes lists: (4)).

Table 2: Secondary endpoints.

## 5. General Study Design and Plan

The study will use retrospectively collected anonymised data from all eligible people contributing to the Optimum Patient Care Research Database (OPCRD)(5) at the date of data extraction. A matched-cohort design will be used for incident (and prevalent) vitiligo related healthcare utilisation, mental health conditions and work impacts. Lifetime risk will be calculated using adapted survival analysis to account for the competing risk of death and will be estimated for the population overall and separately in sociodemographic subgroups of interest.

All adults and adolescents (aged 13+ for disparity objectives 2-5 inclusive) contributing to OPCRD during the study period (January 1, 2004 and December 31, 2020 inclusive). People who have opted out of record data sharing will not be included (approximately 1.8% of the adult population) and have not been uploaded to the OPCRD database.

Cumulative lifetime risk of vitiligo will be estimated (using the method described in the statistical methods below) using cases of incident vitiligo occurring during the observational study period (January 1, 2004 and December 31, 2020 inclusive). A matched-cohort design will be used for incident (and prevalent) vitiligo related mental health conditions, healthcare utilisation and work impacts. For all analyses, the overall result including both adults (aged 18+) and children (aged 13-17) will be published, with stratification by age, sex, deprivation and ethnicity.

## 5.1 Study design

This is a non-interventional study.

## 5.2 Total disease burden; cumulative lifetime risk

A cross sectional design (incidence) will be used to assess the total disease burden of vitiligo, stratified by sociodemographic groups.

# 5.3 Disparities in the impact of vitiligo on mental health, healthcare utilisation and work impact

A matched-cohort design will be used for incident (and prevalent) vitiligo related: Mental health conditions; work impact; healthcare utilisation.

#### 5.4 Data Source and Read codes

The OPCRD(5) is a well-established primary care network in the UK. The database contains complete data on all events and clinical entities coded in UK primary care. These include sociodemographic factors and demographic information, clinical diagnoses, laboratory test results, primary care issued prescriptions, process of care codes (e.g. specialist dermatology reviews), and anthropometric measurements (e.g. BMI), and are coded using the Read coding and Systemized Nomenclature of Medicine – Clinical Terms (SNOMED CT) coding systems.(6)

### 5.5 Data Governance

This study is based wholly on data from the OPCRD (www.opcrd.co.uk) obtained under a limited license from Optimum Patient Care Limited and its execution is approved by recognised experts affiliated to the Respiratory Effectiveness Group.

Data from the OPCRD are available under license for clinical research which is subject to relevant approvals. For additional information visit: <a href="www.opcrd.co.uk">www.opcrd.co.uk</a>.

#### 5.6 Data Extraction

Individual patient data was anonymised at the point of data extraction. All data will remain in anonymised form and will be held on a secure server operated by Momentum Data. The data will not be used for any purposes other than for the research which is described in the respective protocols and which has been approved by the OPCRD ADEPT Committee.

## 5.7 General Study Population

## 5.7.1 Vitiligo Definition

People diagnosed with vitiligo will be identified using diagnostic Read and SNOMED CT codes which are specific to vitiligo. (Appendix 1) A diagnostic algorithm will be used to facilitate robust case identification, identifying anyone with a specific diagnosis code followed by exclusion of anyone with a diagnosis code for an alternative depigmenting

disorder coded within a one-year period (six months before or after their first diagnosis code). The list of alternative depigmenting disorders is shown in Appendix 2.

Incident cases will be defined as people with a first ever diagnosis code of vitiligo during the study period. People with a diagnosis of vitiligo prior to the study period will be excluded. Each case will be assigned an index date at the time of their vitiligo diagnosis.

## 5.7.2 Sociodemographic subgroups

Age, sex, deprivation and ethnicity will comprise the sociodemographic factors used for stratification of the outcome measures.

Age will be stratified into four age categories: 13-17 (adolescents), 18-20, 30-49, 50+.

Ethnicity will be grouped using the standardised definitions of major UK ethnic groups: White, Black, Asian, mixed, and others. (7)

Deprivation will be defined using the national deprivation measure; index of multiple deprivation (IMD) and stratified into quintiles of deprivation according to the national distribution. (8) IMD is calculated at the point of data extraction, using patient postcode (practice postcode where patient postcode is not available).

## 6. Sample Size Calculations

A sample size calculation is only applicable to the incidence of mental health conditions of anxiety and depression in people diagnosed with vitiligo.

Assuming 80% power, a 5% level of statistical significance and a background population prevalence of 15% for anxiety and 10% for depression,(9), our anticipated sample size for vitiligo (n = 8,000) will be sufficient to detect a risk difference of 1.11% in anxiety between those with and without vitiligo, and 1.12% difference in depression between those with and without vitiligo. Sample size calculations were performed in OpenEpi,(10) results are presented using methods of Kelsey.(11)

## 7. Populations to be Analysed

#### 7.1 Inclusion Criteria

People must meet all the following inclusion criteria to be eligible for inclusion in the study:

• The cohort for the endpoint analysis will consist of all adults and adolescents (aged 13+) contributing to OPCRD during the study period.

- The cohort for the lifetime risk analysis will consist of all people contributing to OPCRD during the study period.
- The vitiligo cohort consists of people newly diagnosed with vitiligo at any point during the study period.

#### 7.2 Exclusion Criteria

People meeting any of the following criteria will not be included in the study:

- People with the alternative non-vitiligo diagnoses (other hypopigmenting conditions).
- People with vitiligo diagnosis within 6 months of practice registration.
- People without vitiligo with less than 1 year of follow up within the dataset.
- People over the age of 95 (for those reaching age 95 during the follow up period, follow up was censored at age 95).

People who have opted out of record sharing are not included (approximately 1.8% of the adult population).

## 7.3 Matching Process

For objectives 2-5, controls for each vitiligo case will be identified from the pool of people without a vitiligo diagnosis registered in the OPCRD database at the time of vitiligo diagnosis for the case. Vitiligo cases will be eligible as controls up until the date of their vitiligo diagnosis (at which date their follow-up will be censored if selected as a control).

Each case will be assigned an index date at the time of their vitiligo diagnosis. Corresponding controls assigned to each case will have the same index date.

Each individual with vitiligo will be matched at their index date with up to four unaffected controls. Controls cannot be diagnosed with vitiligo at the date of matching and will require at least one year of follow-up time to minimise the risk of a non-recorded existing diagnosis of vitiligo. Time-updated exact matching will be performed by age, sex, ethnicity and deprivation, selected from the pool of eligible people registered in the same GP practice.

If required, a combination of time-dependent propensity score matching and exact matching will be performed to create a baseline matched dataset.

The matching process is subject to change depending on the feasibility of the mentioned matching process during the initial exploration of the data. The produced baseline matched dataset will be used for all analyses for objective 2-5.

## 8. Statistical Analysis

## 8.1 Statistical Principles

Mean, standard deviation (sd) and any other statistical measures, will be reported to one decimal place. Continuous data will be summarised in the form of means, sd, median, interquartile range (IQR) and range as appropriate. Categorical data will be summarised using the frequencies and proportions. Chi-squared and t-tests will be performed to compare the frequency of dichotomous variables and the values of continuous variables where relevant. 95% CIs will be reported for main effect sizes. Statistical significance will be assessed using p<0.05. Actual p-values will be reported except for p-values less than 3 decimal places which will be reported as "<0.001". P-values >0.1 will be reported to one decimal place, p-values between 0.01 and 0.1 will be reported to 2 decimal places, and p-values between 0.001 and 0.01 will be reported to three decimal places.

The assessment of any associations with baseline characteristics and the outcomes of interest (objectives 2-5) will be assessed using logistic regression (prevalent and incident outcomes), Cox proportional hazards (time to event outcomes) and Poisson regression (repeated event outcomes) models. Three different adjustment sets will be used for each endpoint analysis. These include: an unadjusted model, a sex and age adjusted model, and a multivariable model with an adjustment set of: age, sex, BMI, smoking status, alcohol use, and common comorbidities: type 2 diabetes, hypertension, atrial fibrillation, angina, acute myocardial infarction, stroke, heart failure, chronic liver disease, dementia, rheumatoid arthritis, asthma, chronic obstructive pulmonary disease, chronic kidney disease stages 3-5, malignancy and inflammatory bowel disease.

Assumptions of statistical approaches will be assessed, and transformations used if necessary.

## 8.2 Primary Endpoint Analysis

#### **Objective 1**

Lifetime risk of vitiligo will be calculated for the population as a whole and by sex, ethnicity, and SES. Ethnicity will be grouped using the standardised definitions of major UK ethnic groups: white, black, Asian, mixed, and other.(7) SES will be defined using the national deprivation measure; IMD.(12)

Lifetime risk will be calculated using methods to estimate cumulative lifetime risk recently published in the Lancet, (13, 14) accounting for the competing risk of death. Key outputs will be lifetime risk plots, presenting the cumulative risk of vitiligo against age for the whole population and for sociodemographic subgroups. At a particular age, the cumulative risk estimate can be interpreted as the lifetime risk of vitiligo up until and including the year of age in question. Age of 80 is considered to be the approximate

lifetime expectancy in the UK,(15) and will be the point of comparison at which the lifetime risk of vitiligo will be compared across sociodemographic subgroups.

## 8.3 Secondary Endpoint Analysis

#### **Objective 2**

Anxiety and depression outcomes will be captured if occurring prior to, or within two years of, an individuals' study index date. Binary outcome logistic regression model outputs will be used to compare the burden of anxiety and depression in vitiligo cases compared to matched controls. Furthermore, additional analyses for new onset anxiety and depression outcomes will be conducted, excluding people with a previous record of the respective mental health condition. Anxiety and depression outcomes will be defined by the first occurrence of a relevant code in the primary care record up to two years post index-date. Cox proportional hazards regression will be used to estimate the excess risk of anxiety and depression outcomes in vitiligo cases versus controls. Results will be described as hazard ratios.

#### **Objective 3**

Parasuicide/suicide attempts will be defined by the first occurrence of a relevant code in the primary care record up to two years post index-date. People with a previous record of parasuicide/suicide attempt will be excluded from the calculations. Cox proportional hazards regression will be used to estimate the excess risk of parasuicide/suicide attempts in vitiligo cases versus matched controls. Results will be described as hazard ratios.

Adjustment disorder and sleep disturbance will be defined by the first occurrence of a relevant code in the primary care record up to two years post index-date. People with a previous record of the adjustment disorder will be excluded from the from the adjustment disorder endpoint analysis. Cox proportional hazards regression will be used to estimate the excess risk of the relevant condition in vitiligo cases versus matched controls. Results will be described as hazard ratios.

#### **Objective 4**

Dermatology referral and mental health referral or reviews will be defined by the first occurrence of a relevant code in the primary care record up to two years post index date. Cox proportional hazards regression will be used to estimate the excess risk of these outcomes in vitiligo cases versus matched controls.

For primary care encounters reviews, defined as a rate of encounters within two years after the index date, will be compared using generalised linear models with time-at-risk as an offset. Results will be described as incidence rate ratios.

#### **Objective 5**

Only cases and matched controls aged 18-65 will be considered for this analysis. Work impact outcomes (unemployment and time off work for illness) will be defined by the first occurrence of a relevant code in primary care record up to two years post index date. Cox proportional hazards regression will be used to estimate the excess risk of these outcomes in vitiligo cases versus matched controls. Results will be described as hazard ratios.

## 8.4 Sensitivity Analysis

To evaluate the magnitude of potential bias from including, as matched controls, people who are registered with GP practices but who do not attend their practice, we will also repeat the primary analysis for mental health, healthcare utilisation and work-related outcomes including only matched controls with at least one primary care encounter in the year preceding their index date.

We will also repeat the primary analysis for mental health, healthcare utilisation and work-related outcomes extending the outcome period to four years.

To assess the impact of missing ethnicity data, we will repeat the ethnicity sociodemographic subgroup analysis amending missing ethnicity entries to white.

## 8.5 Missing Data

These studies will use the missing indicator variable method as missing data are considered likely not to be missing at random, meaning multiple imputation approaches will lack validity.

Patients will need to be excluded from analyses based on a matched design if they have incomplete data in the fields (age, sex) required to run the matching process. In similar studies, the exclusion rate due to incomplete data has been very low. (23, 24)

How missing data is handled will be dependent on exploratory and sensitivity analyses and is subject to change.

## 9. Study Limitations

Disparities between sociodemographic subgroups will be interpreted based on the assumption of the primary/secondary outcomes being related to the vitiligo. We have no definite way to identify that every occurrence of an outcome is related to vitiligo in the context of healthcare utilisation and work impact outcomes and therefore causal interpretation is not possible.

This is an ecological study limited to the UK population and may not be generalisable to other populations.

We expect some missing data for the ethnicity variable, this is a limitation of the dataset itself and could result in bias. Necessary sensitivity analyses will be undertaken to circumvent this and limit any impact this could have in interpretation of results in our analysis.

We expect low number of occurrences for the outcomes of referrals for adjustment disorder and parasuicide/suicide, thus reporting of the results for these two endpoints will depend on the sufficiency of numbers available.

## 10. Statistical Software

All statistical analyses will be performed using R version 4.2.3 or higher.

## 11. Ethics

The study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value and rigor and follow generally accepted research practices described in:

- Guidelines for Good Pharmacoepidemiology Practices (GPP). Public Policy Committee, International Society of Pharmacoepidemiology. Pharmacoepidemiology and Drug Safety 2016; 25:2-10.
- Good Practices for Outcomes Research issued by the International Society for Pharmacoeconomics and Outcomes Research (ISPOR)
- Good practices for real-world data studies of treatment and/or comparative effectiveness: Recommendations from the joint ISPOR-ISPE Special Task Force on real-world evidence in health care decision making
- International Ethical Guidelines for Epidemiological Studies issued by the Council for International Organizations of Medical Sciences (CIOMS)
- European Medicines Agency (EMA) European Network of Centres for Pharmacoepidemiology and Pharmacovigilance (ENCePP) Guide on Methodological Standards in Pharmacoepidemiology
- The ENCePP Code of Conduct for scientific independence and transparency in the conduct of pharmacoepidemiological and pharmacovigilance studies
- Good Epidemiological Practice (GEP) guidelines issued by the International Epidemiological Association (IEA).
- Study reporting will be conducted in accordance with the relevant EQUATOR (Enhancing the QUAlity and Transparency Of health Research) guidelines.

The NHS Health Research Authority (NHS HRA) has approved OPCRD for clinical research purposes (REC reference: 20/EM/0148). The protocol for this project was approved by the OPCRD affiliated study approvals committee. The study did not require formal research ethics committee as it used anonymised routinely collected healthcare data, based on outputs from the National Health Service (NHS) Health Research Authority

research decision tool (http://www.hra-decisiontools.org.uk/research/). No patient identifiable information was available to researchers. All patients who chose to opt out of data sharing did not have their data processed. The authors assert that all procedures contributing to this work comply with the ethical standards of the relevant national and institutional committees on human experimentation and with the Helsinki Declaration of 1975, as revised in 2008.

The study will be registered on the clinical trial database (clinicaltrials.gov)

## 12. Acknowledgments

This Study will be based wholly on data from the Optimum Patient Care Research Database (www.opcrd.co.uk) obtained under a limited licence from Optimum Patient Care Limited and its execution is approved by recognised experts affiliated to the Respiratory Effectiveness Group. However, the interpretation and conclusions contained in this report will be those of the author/s alone.

Patients and practices who are members of the OPC network, who allow their data to be shared for surveillance, research, quality improvement, and education. Data access support from the OPCRD team. Statistical input and medical writing from Serhan Bahit (Serhan.bahit@momentumdata.co.uk) and Dr Charlotte Curtis (charlotte.curtis@momentumdata.co.uk) at Momentum Data. Project management support from Emma Jones (emma.jones@momentumdata.co.uk) at Momentum Data.

## 13. References

- 1. Steiner D, Bedin V, Moraes MB, Villas RT, Steiner T. Vitiligo. Anais Brasileiros de Dermatologia. 2004;79:335-51.
- 2. Grimes PE, Miller MM. Vitiligo: Patient stories, self-esteem, and the psychological burden of disease. Int J Womens Dermatol. 2018;4(1):32-7.
- 3. Thompson AR, Eleftheriadou V, Nesnas J. The mental health associations of vitiligo: UK population-based cohort study. BJPsych Open. 2022;8(6):e190.
- 4. Macbeth AE, Holmes S, Harries M, Chiu WS, Tziotzios C, de Lusignan S, et al. The associated burden of mental health conditions in alopecia areata: A population-based study in UK primary care. British Journal of Dermatology.
- 5. Lynam A, Curtis C, Stanley B, Heatley H, Worthington C, Roberts EJ, et al. Data-Resource Profile: United Kingdom Optimum Patient Care Research Database. Pragmat Obs Res. 2023;14:39-49.
- 6. de Lusignan S, Liaw ST, Michalakidis G, Jones S. Defining datasets and creating data dictionaries for quality improvement and research in chronic disease using routinely collected data: an ontology-driven approach. Inform Prim Care. 2011;19(3):127-34.
- 7. Tippu Z, Correa A, Liyanage H, Burleigh D, McGovern A, Van Vlymen J, et al. Ethnicity Recording in Primary Care Computerised Medical Record Systems: An Ontological Approach. J Innov Health Inform. 2017;23(4):920.
- 8. Ministry of Housing, Communities & Local Government, Department for Communities and Local Government. The English Indices of Deprivation. 2015 [updated 23 September 2019. Available from: https://www.gov.uk/government/statistics/english-indices-of-deprivation-2015.
- 9. Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005;62(6):617-27.
- 10. Dean AG, Sullivan KM, Soe MM. OpenEpi: Open Source Epidemiologic Statistics for Public Health [updated 06/04/2013. Available from: <a href="https://www.OpenEpi.com">www.OpenEpi.com</a>.
- 11. Kelsey JL, Whitemore AS, Evans AS, Thompson WD. Methods in Observational Epidemiology. 2nd ed. New York: Oxford University Press; 1996.
- 12. Department for Communities and Local Government. The English Indices of Deprivation. 2015.2015. Available from: <a href="https://www.gov.uk/government/statistics/english-indices-of-deprivation-2015">https://www.gov.uk/government/statistics/english-indices-of-deprivation-2015</a>.
- 13. Gershon AS, Warner L, Cascagnette P, Victor JC, To T. Lifetime risk of developing chronic obstructive pulmonary disease: a longitudinal population study. Lancet (London, England). 2011;378(9795):991-6.
- 14. Rapsomaniki E, Timmis A, George J, Pujades-Rodriguez M, Shah AD, Denaxas S, et al. Blood pressure and incidence of twelve cardiovascular diseases: lifetime risks, healthy life-years lost, and age-specific associations in 1·25 million people. Lancet (London, England). 2014;383(9932):1899-911.
- 15. Minton J, Fletcher E, Ramsay J, Little K, McCartney G. How bad are life expectancy trends across the UK, and what would it take to get back to previous trends? Journal of Epidemiology and Community Health. 2020;74(9):741.

# 14. Appendices

# Appendix 1

Codes to be used to identify cases of vitiligo and important exclusion conditions.

Read and SNOMED codes to be used to identify cases of vitiligo

| Read V2 Code | Term ID | Description |
|---|---|---|
| M2951 | All | Vitiligo |
| M293. | All | Hypopigmentation disorder |
| F4E53 | All | Vitiligo of eyelid |
| M295. | All | Leucoderma |
| M295z | All | Leucoderma NOS |
| Read CTV3 Code | Term ID | Description |
| M2951 | All | Vitiligo |
| M293. | All | Hypopigmentation disorder |
| F4E53 | All | Vitiligo of eyelid |
| M295. | All | Acquired hypomelanosis |
| M295z | All | Leucoderma NOS |
| SNOMED Code | Term ID | Description |
| 56727007 | | Vitiligo (disorder) |
| 87666009 | | Vitiligo of eyelid (disorder) |
| 721539008 | | Vitiligo of eyelid and periocular area (disorder) |
| 403271008 | | Kobner vitiligo (disorder) |
| 403270009 | | Trichrome vitiligo (disorder) |
| 403267005 | | Localised vitiligo (disorder) |
| 403268000 | | Segmental vitiligo (disorder) |
| 402621008 | | Idiopathic vitiligo (disorder) |
| 403269008 | | Generalised vitiligo (disorder) |
| 330931000119106 | | Vitiligo of skin of left eyelid and periocular area (disorder) |
| 330931000119104 | | Vitiligo of skin of right eyelid and periocular area (disorder) |
| 330911000119101 | | Vitiligo of skin of left upper eyelid and periocular area (disorder) |
| 330881000119101 | | Vitiligo of skin of right upper eyelid and periocular area (disorder) |
| 726608002 | | Spastic paraparesis, vitiligo, premature greying, characteristic facies syndrome |
| 23006000 | | Hypopigmentation of skin (disorder) |
| 89031001 | | Hypopigmentation (morphological abnormality) |
| 68210006 | | Hypopigmentation of eyelid |
| 18655006 | | Dipigmentation |
| 23267004 | | Achromia of skin (disorder) |
| 402807009 | | Circumscribed hypomelanosis (disorder) |

Read codes and SNOMED codes to be used to identify alternative depigmenting disorders for exclusion  $% \left( 1\right) =\left( 1\right) \left( 1\right) \left($ 

| Congenital and Genet | tic Hypom | elanoses |
|---|---|---|
| Read V2 Code | Term<br>ID | Description |
| C302A | All | Piebaldism |
| PK5 | All | Tuberous sclerosis |
| PKy54 | All | Waardenburg's syndrome |
| C3029 | All | Hermansky-Pudlak |
| PKy92 | All | Menke's syndrome |
| Read CTV3 Code | Term<br>ID | Description |
| X78Ve | All | Hypomelanosis of Ito |
| XaZqX | All | Piebaldism |
| PK5 | All | Tuberous sclerosis |
| X78E7 | All | Ash leaf spot, tuberous sclerosis |
| X78E8 | All | Shargreen patch |
| X78E9 | All | Adenoma sebaceum |
| X20Ex | All | Hermansky-Pudlak syndrome |
| X20ij | All | Griscelli syndrome with immunodeficiency |
| PKy92 | All | Menkes syndrome |
| SNOMED Code | Term<br>ID | Description |
| 218358001 | | Incontinentia pigmenti achromians syndrome (disorder) |
| 718122005 | | Piebaldism (disorder) |
| 7199000 | | Tuberous sclerosus syndrome (disorder) |
| 254243001 | | Ash leaf spot, tuberous sclerosis (disorder) |
| 36025004 | | Fibrous skin tumor of tuberous sclerosis (disorder) |
| 254244007 | | Shagreen patch (disorder) |
| 9311003 | | Hermansky-Pudlak syndrome (disorder) |
| 37548006 | | Hypopigmentation-immunodeficiency disease (disorder) |
| 59178007 | | Menkes kinky-hair syndrome (disorder) |
| 47434006 | | Waardenburg's syndrome (disorder) |
| 715952000 | | Waardenburg syndrome co-occurrent with Hirschsprung disease (disorder) |
| 773575001 | | Ocular albinism with congenital sensorineural deafness (disorder) |
| 765325002 | | Peripheral demyelinating neuropathy, central dysmyelinating leukodystrophy, Waardenburg syndrome, Hirschsprung disease (disorder) |
| Post-inflammatory H | | oses |
| Read V2 Code | Term<br>ID | Description |
| M2920 | All | Post inflammatory hypopigmentation |
| M170. | All | Lichen planus |

| M1700 | All | Lichen planus actinicus |
|---|---|---|
| M1701 | All | Lichen planus annularis |
| M1702 | All | Lichen planus atrophicus |
| M1702 | All | Lichen planus bullosus |
| M1704 | All | Lichen planus hypertrophicus |
| M1705 | All | Lichen planus linearis |
| M1707 | All | Lichen planus obtusus |
| M1707 | All | Subacute active lichen planus |
| M1708 | All | - |
| M1709 | All | Follicular lichen planus |
| | | Lichen planus NOS |
| M17y0 | All | Lichen ruber moniliforme |
| M1650 | All | Pityriasis alba |
| M2102 | All | Lichen sclerosus and atrophicus |
| K276. | All | Balanitis xerotica obliterans |
| Read CTV3 Code | Term<br>ID | Description |
| Xa0WM | All | Post inflammatory hypopigmentation |
| M170. | All | Lichen planus |
| X507Y | All | Confluent lichen planus |
| X507Z | All | Micropaplular lichen planus |
| X507a | All | Guttate lichen planus |
| X507b | All | Follicular lichen planus |
| M1703 | All | Bullous lichen planus |
| M1701 | All | Annular lichen planus |
| M1704 | All | Hypertrophic lichen planus |
| M1702 | All | Atrophic lichen planus |
| M1705 | All | Linear lichen planus |
| X507c | All | Zosteriform lichen planus |
| M1700 | All | Acintic lichen planus |
| X507d | All | Post inflammatory hyperpigmentation in lichen planus |
| X507e | All | Wickham's striae in lichen planus |
| X507f | All | Lichen planus - lupus erythematosus overlap |
| X507g | All | Lichen planus pemphigoides |
| X507h | All | Site-specific lichen planus |
| X507i | All | Lichen planus of scalp |
| X507j | All | Lichen planus of palms and soles |
| X507k | All | Ulcerative lichen planus of palms and soles |
| X507n | All | Mutilating lichen planus of fingers and toes |
| X507l | All | Lichen planus of nail |
| X507w | All | Genital lichen planus |
| X408F | All | Lichen planus of vuvla |
| X507y | All | Erosive lichen planus of vulva |
| X507z | All | Lichen planus of penis |
| X5080 | All | Lichen planus of glans penis |
| M1707 | All | Lichen planus obtusus |

| M1708 | All | Subacute active lichen planus |
|---|---|---|
| M170z | All | Lichen planus NOS |
| Myu32 | All | [X]Other lichen planus |
| M17y0 | All | Lichen ruber moniliforme |
| M1650 | All | Pityriasis alba |
| M2102 | All | Lichen sclerosus |
| X50FC | All | Genital lichen sclerosus |
| K276. | All | Balanitis xerotica obliterans |
| X50FE | All | Lichen sclerosus of vulva |
| X50FF | All | Extra genital lichen sclerosus |
| X50FG | All | Guttate lichen sclerosus |
| SNOMED Code | Term<br>ID | Description |
| 277787003 | | Post-inflammatory hypopigmentation (disorder) |
| 403272001 | | Post-infective hypomelanosis (disorder) |
| 403276003 | | Acquired hypomelanosis of uncertain etiology (disorder) |
| 4776004 | | Lichen planus (disorder) |
| 263797007 | | Lichen planus-like (qualifier value) |
| 4459000 | | Linear lichen planus (disorder) |
| 6111009 | | Bullous lichen planus (disorder) |
| 238666005 | | Lichen planus of lips (disorder) |
| 201001005 | | Lichen planus obtusus (disorder) |
| 200999007 | | Actinic lichen planus (disorder) |
| 238658001 | | Lichen planus of nail (disorder) |
| 238668006 | | Genital lichen planus (disorder) |
| 201000006 | | Annular lichen planus (disorder) |
| 238647005 | | Guttate lichen planus (disorder) |
| 237112004 | | Lichen planus of vulva (disorder) |
| 400108007 | | Flexural lichen planus (disorder) |
| 238655003 | | Lichen planus of scalp (disorder) |
| 44509000 | | Linear lichen planus (disorder) |
| 25858008 | | Atrophic lichen planus (disorder) |
| 238670002 | | Lichen planus of penis (disorder) |
| 238645002 | | Confluent lichen planus (disorder) |
| 717061002 | | Lichen planus pigmentosus (disorder) |
| 238648000 | | Zosteriform lichen planus (disorder) |
| 238653005 | | Lichen planus pemphigoides (disorder) |
| 68266006 | | Hypertrophic lichen planus (disorder) |
| 238646001 | | Micropapular lichen planus (disorder) |
| 64540004 | | Lichen planopilaris (disorder) |
| 238654004 | | Site-specific lichen planus (disorder) |
| 238652000 | | Lichen planus-lupus erythematosus overlap (disorder) |
| 403198004 | | Lichenoid actinic keratosis (disorder) |
| 723003004 | | Acute eruptive lichen planus (disorder) |
| 238671003 | | Lichen planus of glans penis (disorder) |

| 68266006 | | Hypertrophic lichen planus (disorder) |
|---|---|---|
| 201002003 | | Subacute active lichen planus (disorder) |
| 720493003 | | Annular atrophic lichen planus (disorder) |
| 238651007 | | Wickham's striae in lichen planus (disorder) |
| 201001005 | | Lichen planus obtusus (disorder) |
| 402349005 | | Chronic lichen planus (disorder) |
| 238668006 | | Genital lichen planus (disorder) |
| 238656002 | | Lichen planus of palms and soles (disorder) |
| 402352002 | | Poikiloderma due to lichen planus (disorder) |
| 721171007 | | Hypertrophic lichen planus of vulva (disorder) |
| 402348002 | | Köbner reaction from lichen planus (disorder) |
| 238657006 | | Ulcerative lichen planus of palms and soles (disorder) |
| 238660004 | | Mutilating lichen planus of fingers and toes (disorder) |
| 726476005 | | Lichen planus co-occurrent with onycholysis (disorder) |
| 238649008 | | Post-inflammatory hyperpigmentation in lichen planus (disorder) |
| 402296004 | | Pityriasis alba (disorder) |
| 402298003 | | Diffuse pityriasis alba (disorder) |
| 402297008 | | Localised pityriasis alba (disorder) |
| 25674000 | | Lichen sclerosus et atrophicus (disorder) |
| 402423004 | | Adult lichen sclerosus (disorder) |
| 782666006 | | Lichen sclerosus of anus (disorder) |
| 238934003 | | Guttate lichen sclerosus (disorder) |
| 238932004 | | Genital lichen sclerosus (disorder) |
| 700082001 | | Lichen sclerosus of penis (disorder) |
| 26348009 | | Lichen sclerosus et atrophicus of the vulva (disorder) |
| 402424005 | | Childhood lichen sclerosus (disorder) |
| 403566002 | | Anogenital lichen sclerosus (disorder) |
| 238933009 | | Extragenital lichen sclerosus (disorder) |
| 402714001 | | Lichen sclerosus of male genitalia (disorder) |
| 402715000 | | Lichen sclerosus of female genitalia (disorder) |
| 402422009 | | Bullous extragenital lichen sclerosus (disorder) |
| 721199003 | | Prepubertal lichen sclerosus of vulva (disorder) |
| 403568001 | | Localized extragenital lichen sclerosus (disorder) |
| 402421002 | | Generalized extragenital lichen sclerosus (disorder) |
| 403564004 | | Lichen sclerosus of penis, childhood form (disorder) |
| 111023000 | | Lichen sclerosus et atrophicus, bullous type (disorder) |
| 403565003 | | Vulval lichen sclerosus, childhood form (disorder) |
| 198033005 | | Balanitis xerotica obliterans (disorder) |
| Post Traumatic Leuk | oderma | |
| SNOMED Code | Term<br>ID | Description |
| 402622001 | 12 | Hypomelanosis due to scarring (disorder) |
| 18655006 | | Depigmentation (morphologic abnormality) |
| 23006000 | | Hypopigmentation of skin (disorder) |
| 398656003 | | Acquired hypomelanotic disorder (disorder) |
| <u> </u> | l | 1 |

| Para-Malignant Hypor | melanoses | |
|---|---|---|
| Read V2 Code | Term<br>ID | Description |
| B621. | All | Mycosis fungoides |
| B6210 | All | Mycosis fungoides of unspecified site |
| B6211 | All | Mycosis fungoides of lymph nodes of head, face and neck |
| B6212 | All | Mycosis fungoides of intrathoracic lymph nodes |
| B6213 | All | Mycosis fungoides of intra-abdominal lymph nodes |
| B6214 | All | Mycosis fungoides of lymph nodes of axilla and upper limb |
| B6215 | All | Mycosis fungoides of lymph nodes of inguinal region and leg |
| B6216 | All | Mycosis fungoides of intrapelvic lymph nodes |
| B6217 | All | Mycosis fungoides of spleen |
| B6218 | All | Mycosis fungoides of lymph nodes of multiple sites |
| B621z | All | Mycosis fungoides NOS |
| BBI | All | [M]Mycosis fungoides |
| BBIO. | All | [M]Mycosis fungoides |
| BBI1. | All | [M]Sezary's disease |
| BBIz. | All | [M]Mycosis fungoides NOS |
| B62xX | All | 0th and unspecif peripheral & cutaneous T-cell lymphomas |
| B62E7 | All | Subcutaneous panniculitis like T-cell lymphoma |
| BBmD. | All | [M]Cutaneous lymphoma |
| B622. | All | Sezary's disease |
| B6220 | All | Sezary's disease of unspecified site |
| B6221 | All | Sezary's disease of lymph nodes of head, face and neck |
| B6222 | All | Sezary's disease of intrathoracic lymph nodes |
| B6223 | All | Sezary's disease of intra-abdominal lymph nodes |
| B6224 | All | Sezary's disease of lymph nodes of axilla and upper limb |
| B6225 | All | Sezary's disease of lymph nodes of inguinal region and leg |
| B6226 | All | Sezary's disease of intrapelvic lymph nodes |
| B6227 | All | Sezary's disease of spleen |
| B6228 | All | Sezary's disease of lymph nodes of multiple sites |
| B622z | All | Sezary's disease NOS |
| BBEA. | All | Amelanotic melanoma |
| Read CTV3 Code | Term<br>ID | Description |
| B621. | All | Mycosis fungoides |
| XaQbT | All | Poikiloderma vasculare atrophicans |
| X78hm | All | Mycosis fungoides of skin |
| B6210 | All | Mycosis fungoides of unspecified site |
| B6211 | All | Mycosis fungoides of lymph nodes of head, face and neck |
| B6212 | All | Mycosis fungoides of intrathoracic lymph nodes |
| B6213 | All | Mycosis fungoides of intra-abdominal lymph nodes |
| B6214 | All | Mycosis fungoides of lymph nodes of axilla and upper limb |
| B6215 | All | Mycosis fungoides of lymph nodes of inguinal region and leg |
| B6216 | All | Mycosis fungoides of intrapelvic lymph nodes |

| B6217 | All | Mycosis fungoides of spleen |
|---|---|---|
| B6218 | All | Mycosis fungoides of lymph nodes of multiple sites |
| B621z | All | Mycosis fungoides NOS |
| B622. | All | Sezary's disease |
| B6220 | All | Sezary's disease of unspecified site |
| B6221 | All | Sezary's disease of lymph nodes of head, face and neck |
| B6222 | All | Sezary's disease of intrathoracic lymph nodes |
| B6223 | All | Sezary's disease of intra-abdominal lymph nodes |
| B6224 | All | Sezary's disease of lymph nodes of axilla and upper limb |
| B6225 | All | Sezary's disease of lymph nodes of inguinal region and leg |
| B6226 | All | Sezary's disease of intrapelvic lymph nodes |
| B6227 | All | Sezary's disease of spleen |
| B6228 | All | Sezary's disease of lymph nodes of multiple sites |
| B622z | All | Sezary's disease NOS |
| X78hn | All | Sezary's disease of skin |
| X78hl | All | Cutaneous lymphoma |
| XaYin | All | Cutaneous follicle centre lymphoma |
| Xa0Sz | All | Cutaneous/peripheral T-cell lymphoma |
| XaYjf | All | Subcutaneous panniculitis like T-cell lymphoma |
| ByuDD | All | [X]0th and unspecif peripheral & cutaneous T-cell lymphomas |
| XaYjl | All | Primary cutaneous CD30 antigen positive large T-cell lymphoma |
| 1M1 J1 | | |
| XaOCE | All | Amelanotic malignant melanoma of skin |
| | All Term ID | Amelanotic malignant melanoma of skin Description |
| XaOCE | Term | - |
| XaOCE SNOMED Code | Term | Description |
| XaOCE SNOMED Code 90120004 | Term | Description Mycosis fungoides (morphologic abnormality) |
| XaOCE SNOMED Code 90120004 118618005 | Term | Description Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) |
| XaOCE SNOMED Code 90120004 118618005 765328000 | Term | Description Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) |
| XaOCE SNOMED Code 90120004 118618005 765328000 404115006 | Term | Description Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) |
| XaOCE SNOMED Code 90120004 118618005 765328000 404115006 94714002 | Term | Description Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) |
| XaOCE SNOMED Code 90120004 118618005 765328000 404115006 94714002 404117003 | Term | Description Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) |
| XaOCE SNOMED Code 90120004 118618005 765328000 404115006 94714002 404117003 681291000119105 | Term | Description Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) |
| XaOCE SNOMED Code 90120004 118618005 765328000 404115006 94714002 404117003 681291000119105 418628003 | Term | Description Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) |
| XaOCE SNOMED Code 90120004 118618005 765328000 404115006 94714002 404117003 681291000119105 418628003 404113004 | Term | Description Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) |
| XaOCE SNOMED Code 90120004 118618005 765328000 404115006 94714002 404117003 681291000119105 418628003 404113004 404118008 | Term | Description Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) |
| XaOCE SNOMED Code 90120004 118618005 765328000 404115006 94714002 404117003 681291000119105 418628003 404113004 404118008 404112009 | Term | Description Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) Granulomatous mycosis fungoides (disorder) |
| XaOCE SNOMED Code 90120004 118618005 765328000 404115006 94714002 404117003 681291000119105 418628003 404113004 404118008 404112009 404114005 | Term | Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) Granulomatous mycosis fungoides (disorder) Erythrodermic mycosis fungoides (disorder) |
| XaOCE SNOMED Code 90120004 118618005 765328000 404115006 94714002 404117003 681291000119105 418628003 404113004 404118008 404112009 404114005 404110001 | Term | Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) Granulomatous mycosis fungoides (disorder) Erythrodermic mycosis fungoides (disorder) Hypomelanocytic mycosis fungoides (disorder) |
| XaOCE SNOMED Code 90120004 118618005 765328000 404115006 94714002 404117003 681291000119105 418628003 404113004 404118008 404112009 404114005 404110001 404109006 | Term | Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) Granulomatous mycosis fungoides (disorder) Erythrodermic mycosis fungoides (disorder) Hypomelanocytic mycosis fungoides (disorder) Folliculotropic mycosis fungoides (disorder) |
| XaOCE SNOMED Code 90120004 118618005 765328000 404115006 94714002 404117003 681291000119105 418628003 404113004 404118008 404112009 404114005 404110001 404109006 404108003 | Term | Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) Granulomatous mycosis fungoides (disorder) Erythrodermic mycosis fungoides (disorder) Hypomelanocytic mycosis fungoides (disorder) Folliculotropic mycosis fungoides (disorder) Pokilodermatous mycosis fungoides (disorder) |
| XaOCE SNOMED Code 90120004 118618005 765328000 404115006 94714002 404117003 681291000119105 418628003 404113004 404118008 404112009 404114005 404109006 404108003 404107008 | Term | Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) Granulomatous mycosis fungoides (disorder) Erythrodermic mycosis fungoides (disorder) Hypomelanocytic mycosis fungoides (disorder) Folliculotropic mycosis fungoides (disorder) Pokilodermatous mycosis fungoides (disorder) Patch/plaque stage mycosis fungoides (disorder) |
| XaOCE SNOMED Code 90120004 118618005 765328000 404115006 94714002 404117003 681291000119105 418628003 404113004 404118008 404112009 404114005 404110001 404109006 404108003 404107008 404116007 | Term | Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) Granulomatous mycosis fungoides (disorder) Erythrodermic mycosis fungoides (disorder) Hypomelanocytic mycosis fungoides (disorder) Folliculotropic mycosis fungoides (disorder) Pokilodermatous mycosis fungoides (disorder) Patch/plaque stage mycosis fungoides (disorder) Mycosis fungoides with systemic infiltration (disorder) |
| XaOCE SNOMED Code 90120004 118618005 765328000 404115006 94714002 404117003 681291000119105 418628003 404113004 404118008 404112009 404114005 404109006 404109006 404108003 404107008 404116007 94708009 | Term | Mycosis fungoides (morphologic abnormality) Mycosis fungoides (disorder) Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) Granulomatous mycosis fungoides (disorder) Erythrodermic mycosis fungoides (disorder) Hypomelanocytic mycosis fungoides (disorder) Folliculotropic mycosis fungoides (disorder) Pokilodermatous mycosis fungoides (disorder) Patch/plaque stage mycosis fungoides (disorder) Mycosis fungoides with systemic infiltration (disorder) Mycosis fungoides of intrapelvic lymph nodes (disorder) |

| 404104001 | Lymphomatoid papulosis type B mycosis fungoides-like (disorder) |
|---|---|
| 94715001 | Mycosis fungoides of extranodal AND/OR solid organ site (disorder) |
| 94709001 | Mycosis fungoides of intrathoracic lymph nodes (disorder) |
| 94711005 | Mycosis fungoides of lymph nodes of head, face AND/OR neck (disorder) |
| 94710006 | Mycosis fungoides of lymph nodes of axilla AND/OR upper limb (disorder) |
| 188627002 | Mycosis fungoides of lymph nodes of multiple sites (disorder) |
| 94712003 | Mycosis fungoides of lymph nodes of inguinal region AND/OR lower limb (disorder) |
| 28054005 | Cutaneous T-cell lymphoma, no International Classification of Diseases for oncology subtype (morphologic abnormality) |
| 40012207 | Primary cutaneous T-cell lymphoma (disorder) |
| 277613000 | Cutaneous/peripheral T-cell lymphoma (disorder) |
| 404128004 | CD-30 negative cutanoeus T-cell lymphoma (disorder) |
| 419283005 | Primary cutaneous T-cell lymphoma - category (morphologic abnormality) |
| 128804002 | Primary cutaneous CD30 antigen positive T-cell lymphoproliferative disorder (morphologic abnormality) |
| 450908002 | Primary cutaneous gamma-delta T-cell lymphoma (morphologic abnormality) |
| 122571000119106 | History of primary cutaneous T-cell lymphoma (situation) |
| 419018000 | Primary cutaneous large T-cell lymphoma - category (morphologic abnormality) |
| 402880009 | Primary cutaneous large T-cell lymphoma (disorder) |
| 404133000 | Subcutaneous panniculitic cutaneous T-cell lymphoma (disorder) |
| 404128004 | CD-30 negative cutaneous T-cell lymphoma (disorder) |
| 787198005 | Primary cutaneous acral CD8 positive T-cell lymphoma (morphologic abnormality) |
| 397352006 | Primary cutaneous anaplastic large T-cell lymphoma, CD30-positive (morphologic abnormality) |
| 733627006 | Primary cutaneous gamma-delta-positive T-cell lymphoma (disorder) |
| 404129007 | CD-30 negative anaplastic large T-cell cutaneous lymphoma (disorder) |
| 122571000119106 | History of malignant cutaneous T-cell lymphoma (situation) |
| 404130002 | CD-30 negative pleomorphic large T-cell cutaneous lymphoma (disorder) |
| 404126000 | CD-30 positive pleomorphic large T-cell cutaneous lymphoma (disorder) |
| 419283005 | Primary cutaneous T-cell lymphoma - category (morphologic abnormality) |
| 450908002 | Primary cutaneous gamma-delta T-cell lymphoma - category (morphologic abnormality) |
| 765136002 | Primary cutaneous CD8 positive aggressicve epidermotropic cytotoxic T-cell lymphoma (disorder) |
| 128875000 | Primary cutaneous CD30 antigen positive large T-cell lymphoma (disorder) |
| 733895005 | Primary cutaneous CD8 positive aggressicve epidermotropic cytotoxic T-cell lymphoma (morphologic abnormality) |

| | Primary cutaneous T-cell lymphoma, large cell, CD30-negative |
|---|---|
| | (morphological abnormality) |
| | Sezary's disease (disorder) |
| | Sezary's disease (morphologic abnormality) |
| | Sezary disease of skin (disorder) |
| | Sezary's disase of spleen (disorder) |
| | Sezary's disase of intra-abdominal lymph nodes (disorder) |
| | Sezary's disase of intrapelvic lymph nodes (disorder) |
| | Sezary's disase of intrathoracic lymph nodes (disorder) |
| | Sezary disease of lymph nodes of multiple sites (disorder) |
| | Sézary's disease of extranodal AND/OR solid organ site (disorder) |
| | Sézary's disease of lymph nodes of axilla and upper limb (disorder) |
| | Sézary's disease of lymph nodes of head, face AND/OR neck (disorder) |
| | Sézary's disease of lymph nodes of inguinal region and lower limb (disorder) |
| | Sézary's disease of lymph nodes of inguinal region AND/OR lower limb (disorder) |
| | Primary cutaneous lymphoma (morphologic abnormality) |
| | Tumour and germline whole genome sequencing for anaplastic lymphoma kinase negative anaplastic large cell lymphoma including |
| | primary cutaneous subtypes (procedure) |
| | Hypomelanosis surrounding malignant melanoma (disorder) |
| | Metastatic malignant melanoma with diffuse hypermelanosis (disorder) |
| | Amelanotic malignant melanoma of skin (disorder) |
| | Amelanotic melanoma (morphologic abnormality) |
| | Hypomelanotic mycosis fungoides (disorder) |
| | Hypomelanosis surrounding melanocytic neoplasm (disorder) |
| nduced hy | pomelanoses |
| Term<br>ID | Description |
| All | Hypopigmentation |
| Term<br>ID | Description |
| All | Occupational vitiligo |
| All | Chemically-induced hypomelanosis |
| All | Drug-induced hypomelanosis |
| All | Chemically-induced hypomelanosis |
| All | Leucoderma aestivale |
| All | Acquired hypomelanosis |
| Term<br>ID | Description |
| | Occupational vitiligo (disorder) |
| | Chemically-induced hypomelanosis (disorder) |
| | Chemicany-mudeed hypometanosis (disorder) |
| | Term ID All Term ID All All All All All All All Term |

| 403807001 | | Phylloid hypomelanosis (disorder) |
|---|---|---|
| 398656003 | | Acquired hypomelanotic disorder (disorder) |
| 238999005 | | Drug-induced hypomelanosis (disorder) |
| 403698000 | | Laser-induced hypopigmentation (disorder) |
| 402622001 | | Hypomelanosis due to scarring (disorder) |
| 280962005 | | Chemically-induced hypomelanosis (disorder) |
| 403692004 | | Hypomelanosis due to cryotherapy (disorder) |
| 403744007 | | Arsenic-induced "rain-drop" hypomelanosis (disorder) |
| 403698000 | | Laser-induced hypopigmentation (disorder) |
| 201290009 | | Leukoderma estivale (disorder) |
| Para-infectious hypo | <br>nigmentat | 1 |
| Read V2 Code | Term<br>ID | Description |
| AB10. | All | Pityriasis versicolor |
| Read CTV3 Code | Term<br>ID | Description |
| AB10. | All | Pityriasis versicolor |
| SNOMED Code | Term<br>ID | Description |
| 56454009 | | Pityriasis versicolor (disorder) |
| 18097004 | | Malassezia (organism) |
| 721794002 | | Infection caused by Malassezia (disorder) |
| 402133004 | | Malassezia infection of the skin (disorder) |
| 29619007 | | Malassezia furfur (organism) |
| Others (including Mela | | Malassezia furfur (organism) hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) |
| Others (including Mela | | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, |
| Others (including Mela<br>Progressive macular h | ypomelano<br><b>Term</b> | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) |
| Others (including Mela<br>Progressive macular hy<br>Read V2 Code | ypomelano<br>Term<br>ID | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) Description |
| Others (including Mela<br>Progressive macular h<br>Read V2 Code<br>M290. | ypomelano Term ID All | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) Description Melasma |
| Others (including Mela<br>Progressive macular hy<br>Read V2 Code<br>M290.<br>M2900 | ypomelano Term ID All All | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) Description Melasma Chloasma bronzinum |
| Others (including Mela<br>Progressive macular hy<br>Read V2 Code<br>M290.<br>M2900<br>M2901 | Term ID All All All | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) Description Melasma Chloasma bronzinum Chloasma cachecticorum |
| Others (including Mela<br>Progressive macular hy<br>Read V2 Code<br>M290.<br>M2900<br>M2901<br>M2902 | Term ID All All All All | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) Description Melasma Chloasma bronzinum Chloasma cachecticorum Chloasma caloricum |
| Others (including Mela<br>Progressive macular hy<br>Read V2 Code<br>M290.<br>M2900<br>M2901<br>M2902<br>M2903 | ypomelano Term ID All All All All All | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) Description Melasma Chloasma bronzinum Chloasma cachecticorum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum |
| Others (including Mela<br>Progressive macular hy<br>Read V2 Code<br>M290.<br>M2900<br>M2901<br>M2902<br>M2903<br>M2903 | Term ID All All All All All All | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) Description Melasma Chloasma bronzinum Chloasma cachecticorum Chloasma gravidarum Chloasma gravidarum |
| Others (including Mela<br>Progressive macular hy<br>Read V2 Code<br>M290.<br>M2900<br>M2901<br>M2902<br>M2903<br>M2903<br>M2903 | ypomelano Term ID All | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) Description Melasma Chloasma bronzinum Chloasma cachecticorum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum |
| Others (including Mela<br>Progressive macular hy<br>Read V2 Code<br>M290.<br>M2900<br>M2901<br>M2902<br>M2903<br>M2903<br>M2903<br>M2903<br>M2903 | Term ID All Al | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) Description Melasma Chloasma bronzinum Chloasma cachecticorum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma nos |
| Others (including Mela<br>Progressive macular hy<br>Read V2 Code<br>M290.<br>M2900<br>M2901<br>M2902<br>M2903<br>M2903<br>M2903<br>M2903<br>M2903<br>M2903 | ypomelano Term ID All Al | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) Description Melasma Chloasma bronzinum Chloasma cachecticorum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma hoos Morphoea Linear Morphoea Circumscribed scleroderma |
| Others (including Mela<br>Progressive macular hy<br>Read V2 Code<br>M290.<br>M2900<br>M2901<br>M2902<br>M2903<br>M2903<br>M2903<br>M2903<br>M2903<br>M2903<br>M2904 | Term ID All All All All All All All A | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) Description Melasma Chloasma bronzinum Chloasma cachecticorum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma MOS Morphoea Linear Morphoea |
| Others (including Mela<br>Progressive macular hy<br>Read V2 Code M290. M2900 M2901 M2902 M2903 M2903 M2903 M2903 M2903 M2904 M2104 M210. | Term ID All Al | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) Description Melasma Chloasma bronzinum Chloasma cachecticorum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma hoos Morphoea Linear Morphoea Circumscribed scleroderma |
| Others (including Mela<br>Progressive macular hy<br>Read V2 Code M290. M2900 M2901 M2902 M2903 M2903 M2903 M2903 M2903 M2904 M2100 M2104 M2100 | Term ID All All All All All All All A | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) Description Melasma Chloasma bronzinum Chloasma cachecticorum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma MOS Morphoea Linear Morphoea Circumscribed scleroderma Unspecified circumscribed scleroderma |
| Others (including Mela<br>Progressive macular hy<br>Read V2 Code M290. M2900 M2901 M2902 M2903 M2903 M2903 M2903 M2903 M2100 M2100 M2100 M2101 | Term ID All Al | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) Description Melasma Chloasma bronzinum Chloasma cachecticorum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma pravidarum Chloasma gravidarum Chloasma NOS Morphoea Linear Morphoea Circumscribed scleroderma Unspecified circumscribed scleroderma Localised dermatosclerosis |
| Others (including Mela<br>Progressive macular hy<br>Read V2 Code M290. M2900 M2901 M2902 M2903 M2903 M2903 M2903 M2903 M2104 M2100 M2100 M2101 M2100 | Term ID All All All All All All All A | hoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, sis, Nevus depigmentosus, Cutaneous sarcoidosis) Description Melasma Chloasma bronzinum Chloasma cachecticorum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma gravidarum Chloasma nos Morphoea Linear Morphoea Circumscribed scleroderma Unspecified circumscribed scleroderma Localised dermatosclerosis Circumscribed scleroderma NOS |

| AD53. | All | Sarcoidosis of skin |
|----------------|------------|---------------------------------------|
| Read CTV3 Code | Term<br>ID | Description |
| M290. | All | Melasma |
| Xa1aM | All | Drug-induced melasma |
| M2900 | All | Chloasma bronzinum |
| M2901 | All | Chloasma cachecticorum |
| M2902 | All | Chloasma caloricum |
| M2904 | All | Chloasma hepaticum |
| M2905 | All | Chloasma toxicum |
| M2906 | All | Chloasma traumaticum |
| M290z | All | Chloasma NOS |
| M2903 | All | Melasma of pregnancy |
| Xa1aM | All | Drug-induced melasma |
| M2103 | All | Morphoea |
| X7053 | All | Generalised morphoea |
| M2101 | All | Localised morphoea |
| M2100 | All | Unspecified circumscribed scleroderma |
| M210z | All | Circumscribed scleroderma NOS |
| X7055 | All | Linear morphoea |
| PH322 | All | Xeroderma pigmentosum |
| X78Cz | All | Xeroderma pigmentosum group A |
| X78D0 | All | Xeroderma pigmentosum group B |
| X78D1 | All | Xeroderma pigmentosum group C |
| X78D2 | All | Xeroderma pigmentosum group D |
| X78D3 | All | Xeroderma pigmentosum group E |
| X78D4 | All | Xeroderma pigmentosum group F |
| X78D5 | All | Xeroderma pigmentosum group G |
| X78D6 | All | Xeroderma pigmentosum XP variant |
| X78D7 | All | De Sanctis-Cacchione syndrome |
| X78D8 | All | Xerodermoid, pigmented |
| X50lw | All | Symmetrical progressive leucopathy |
| X20GW | All | Cutaneous sarcoid |
| X20GX | All | Orofacial sarcoid |
| X20GY | All | Lupus pernio |
| X5089 | All | Acute skin sarcoidosis |
| X508A | All | Sarcoidosis-induced erythema nodosum |
| X508B | All | Lofgrens syndrome |
| X508C | All | Maculopapular sarcoidosis |
| X508D | All | Chronic skin sarcoidosis |
| X508E | All | Sarcoidosis in scar |
| X508F | All | Papular sarcoidosis |
| X508G | All | Lichenoid sarcoidosis |
| X508H | All | Nodular sarcoidosis |
| X508I | All | Angiolupoid sarcoidosis |
| | * **** | 1 B-o-upora our coracoro |

| X00YQ | All | Sarcoid skin of eyelid |
|---|---|---|
| X20G5 | All | Sarcoid dactylitis |
| X50Dy | All | Subacute nodular migratory panniculitis |
| X50Dz | All | Subcutaneous lipogranulomatosis |
| SNOMED Code | Term<br>ID | Description |
| 36209000 | | Melasma |
| 201274009 | | Chloasma bronzinum (disorder) |
| 201275005 | | Chloasma cachecticorum (disorder) |
| 201276006 | | Chloasma caloricum (disorder) |
| 201277002 | | Chloasma hepaticum (disorder) |
| 201278007 | | Chloasma toxicum (disorder) |
| 280955001 | | Drug-induced melasma (disorder) |
| 79840007 | | Idiopathic chloasma (disorder) |
| 111208003 | | Melasma gravidarum (disorder) |
| 54397000 | | Symptomatic chloasma (disorder) |
| 201279004 | | Chloasma traumaticum (disorder) |
| 201049004 | | Morphea (disorder) |
| 128458002 | Plaque morphea (disorder) | |
| 22784002 | Linear scleroderma (disorder) | |
| 403521006 | Guttate morphea (disorder) | |
| 201048007 | | Localised morphea (disorder) |
| 7513007 | | Generalized morphea (disorder) |
| 403522004 | | Subcutaneous morphea (disorder) |
| 51156002 | | Coup de sabre scleroderma (disorder) |
| 403523009 | | Disabling pansclerotic morphea of children (disorder) |
| 128460000 | | Diffuse cutaneous scleroderma (disorder) |
| 403524003 | | Scleroderma-like secondary cutaneous sclerosis (disorder) |
| 1717003 | | Idiopathic guttate hypomelanosis (disorder) |
| 711154007 | | Guttate hypopigmentation and punctate palmoplantar keratoderma with or without ectopic calcification (disorder) |
| 44600005 | | Xeroderma pigmentosum (disorder) |
| 56048001 | | Xeroderma pigmentosum, group E (disorder) |
| 25784009 | | Xeroderma pigmentosum, group C (disorder) |
| 36454001 | | Xeroderma pigmentosum, group G (disorder) |
| 1073003 | | Xeroderma pigmentosum, group B (disorder) |
| 68637004 | | Xeroderma pigmentosum, group D (disorder) |
| 42530008 | | Xeroderma pigmentosum, group F (disorder) |
| 43477006 | | Xeroderma pigmentosum, group A (disorder) |
| 73663008 | | Neurologic xeroderma pigmentosum (disorder) |
| 88877002 | | Xeroderma pigmentosum, variant form (disorder) |
| 7806002 | | Non-neurologic xeroderma pigmentosum (disorder) |
| 719819004 | | Xeroderma pigmentosum and Cockayne syndrome complex (disorder) |
| 239083007 | | Symmetrical progressive leucopathy (disorder) |

| 763368004 | Familial progressive hyper and hypopigmentation of skin (disorder) |
|---|---|
| 403541001 | Nevus depigmentosus |
| 112680001 | Naevus depigmentosus |
| 55941000 | Cutaneous sarcoidosis (disorder) |
| 238680003 | Papular sarcoidosis (disorder) |
| 238679001 | Sarcoidosis in scar (disorder) |
| 402369000 | Atrophic sarcoidosis (disorder) |
| 402371000 | Verrucous sarcoidosis (disorder) |
| 238681004 | Lichenoid sarcoidosis (disorder) |
| 238674006 | Acute skin sarcoidosis (disorder) |
| 402370004 | Ulcerative sarcoidosis (disorder) |
| 58870009 | Sarcoidosis, anular type (disorder) |
| 54515008 | Sarcoidosis, plaque type (disorder) |
| 80941006 | Subcutaneous sarcoidosis (disorder) |
| 870334009 | Palmoplantar sarcoidosis (disorder) |
| 238678009 | Chronic skin sarcoidosis (disorder) |
| 238677004 | Maculopapular sarcoidosis (disorder) |
| 402368008 | Ichthyosiform sarcoidosis (disorder) |
| 402373002 | Hypomelanotic sarcoidosis (disorder) |
| 9529007 | Sarcoidosis, erythrodermic type (disorder) |
| 72470008 | Sarcoidosis, lupus pernio type (disorder) |
| 402372007 | Subcutaneous nodular sarcoidosis (disorder) |
| 238675007 | Sarcoidosis-induced erythema nodosum (disorder) |
| 238676008 | Lofgrens syndrome (disorder) |
| 31541009 | Lupus pernio of Besnier |
| 231799005 | Sarcoid skin of eyelid (disorder) |

# Appendix 2

Potential differential diagnoses for vitiligo which will be used as exclusion criteria if they appear as diagnoses in the medical record within six months of the initial diagnosis of vitiligo (six months before or after the vitiligo diagnosis). \*As these conditions are extremely uncommon in the UK they will not be used in the exclusion process. Codes for these conditions are listed in Appendix 1.

| Condition group | Conditions/causes included |
|---|---|
| Congenital and genetic hypomelanoses | Piebaldism |
| | Tuberous sclerosis |
| | Hypomelanosis of Ito |
| | Waardenburg syndrome |
| | Hermanski-Pudlak syndrome |
| | Griscelli syndrome |
| | Menkes syndrome |
| Post-inflammatory hypomelanoses | Post-inflammatory leukoderma including after |
| | Atopic eczema or Psoriasis |
| | Lichen planus |
| | Pityriasis alba |
| | Lichen sclerosus |
| Post traumatic leukoderma | Post traumatic leukoderma |
| Para-malignant hypomelanoses | Cutaneous T-cell lymphoma (mycosis fungoides) |
| | Melanoma associated depigmentation |
| Occupational/drug induced | Occupational vitiligo |
| hypomelanoses | Other induced hypomelanoses |
| Para-infectious hypopigmentation | Pityriasis versicolor (or tinea versicolor) |
| | Leprosy* |
| | Leishmaniasis* |
| Others | Melasma |
| | Morphoea |
| | Idiopathic guttate hypomelanosis |
| | Xeroderma pigmentosum |
| | Progressive macular hypomelanosis |
| | Nevus depigmentosus |
| | Cutaneous sarcoidosis |